CLINICAL TRIAL: NCT00504829
Title: A 12-Week, Multi-Center, Double-Blind, Randomized, Parallel-Group Study, Followed by a 12 Month Extension Study, of the Efficacy and Safety of LCP-AtorFen in Subjects With Dyslipidemia
Brief Title: Study of Atorvastatin/Fenofibrate (LCP-AtorFen) Combination Therapy in Dyslipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCP-AtorFen-2001
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Dyslipidemia
Keywords: LCP-AtorFen; Non-HDL cholesterol; Triglycerides; HDL cholesterol; LDL cholesterol; Atorvastatin; Fenofibrate
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LCP-AtorFen (Experimental): LCP-AtorFen 40/100mg fixed-dose combination tablet of 40mg atorvastatin and 145mg fenofibrate for treatment of mixed dyslipidemia
  Interventions: Drug: LCP-AtorFen
- atorvastatin (Active Comparator): atorvastatin 40mg tablet (Lipitor), as an adjunct to diet and exercise for treatment of mixed dyslipidemia
  Interventions: Drug: atorvastatin
- fenofibrate (Active Comparator): fenofibrate 145mg tablet (Tricor), as an adjunct to diet and exercise for treatment of mixed dyslipidemia
  Interventions: Drug: fenofibrate

INTERVENTIONS:
Drug: LCP-AtorFen — 40mg atorvastatin combined with 100mg fenofibrate in a tablet for once daily treatment of dyslipidemia and mixed dyslipidemia
  Arms: LCP-AtorFen
Drug: atorvastatin — dyslipidemia and mixed dyslipidemia
  Other Names: Lipitor
  Arms: atorvastatin
Drug: fenofibrate — dyslipidemia and mixed dyslipidemia
  Other Names: Tricor
  Arms: fenofibrate

SUMMARY:
The current study is designed to test the efficacy, safety and tolerability of LCP-AtorFen, a combination of atorvastatin and fenofibrate.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, 12 week study with a 52-week open-label follow-up to evaluate the safety and efficacy of LCP-AtorFen (the combination of atorvastatin and fenofibrate) in the treatment of hyperlipidemia.

After a wash-out phase, eligible patients will be randomized on a 1:1:1 ratio to either LCP-AtorFen, atorvastatin or fenofibrate for 12 weeks. After the completion of the 12-week phase, all eligible patients will be offered to receive open-label LCP-AtorFen for another 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of dyslipidemia (non-HDL-C >130 mg/dL and Triglycerides > or equal to 150 mg/dL and < or equal to 500 mg/dL).
2. Subject may be currently on a statin or other lipid-lowering therapy but must be willing and able to washout for 8 weeks if on a fibrate or high-dose niacin, 6 weeks if on a statin or low-dose niacin per day, or 4 weeks if on a bile acid sequestrant, ezetimibe, or >1000 mg of fish oil per day.
3. Other inclusion criteria might apply

Exclusion Criteria:

1. TGs > 500 mg/dL.
2. History of coronary heart disease (CHD), transient ischemic attacks, stroke or revascularization procedure in the six months prior.
3. Presence of an aortic aneurysm or resection of an aortic aneurysm within six months.
4. Poorly controlled diabetes mellitus (glycosylated hemoglobin >8.0% )or diabetes mellitus requiring insulin therapy.
5. Known lipoprotein lipase impairment or deficiency or Apo C-II deficiency or familial dysbetalipoproteinemia.
6. History of pancreatitis.
7. Known allergy or sensitivity to statins or fibrates.
8. Poorly controlled hypertension.
9. Other exclusion criteria might apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2007-07; Primary Completion 2008-02 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Geohas, MD, Principal Investigator — Radiant Research; Dennis McCluskey, MD, Study Director — Radiant Research; Harry Geisberg, MD, Study Director — Radiant Research; Chivers Woodruff, Jr, MD, Study Director — Radiant Research; Michael Noss, MD, Study Director — Radiant Research; Michele Reynolds, MD, Study Director — Radiant Research; James Zavoral, MD, Study Director — Radiant Research; Randall Severance, MD, Study Director — Radiant Research; Stephen Halpern, MD, Study Director — Radiant Research; Linda Murray, MD, Study Director — Radiant Research; Wayne Larson, MD, Study Director — Radiant Research; Timothy Howards, MD, Study Director — Medical Affiliated Research Center, Inc.; Cynthia Strout, MD, Study Director — Coastal Carolina Research Center; Mark Kipnes, MD, Study Director — Diabetes and Glandular Research Center, Inc.
Locations (1):
- Radiant Research, 515 N State Street, Suite 2700, Chicago, Illinois, United States

REFERENCES:
- [Derived] Davidson MH, Rooney MW, Drucker J, Eugene Griffin H, Oosman S, Beckert M; LCP-AtorFen Investigators. Efficacy and tolerability of atorvastatin/fenofibrate fixed-dose combination tablet compared with atorvastatin and fenofibrate monotherapies in patients with dyslipidemia: a 12-week, multicenter, double-blind, randomized, parallel-group study. Clin Ther. 2009 Dec;31(12):2824-38. doi: 10.1016/j.clinthera.2009.12.007. PMID 20110022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited from a combination of sources: advertising, clinical databases, clinical referrals, and the general subject population.
Pre-assignment Details: The washout period for subjects on lipid-lowering therapy will be 4 to 8 weeks, depending on their regimen.
Groups:
- LCP-AtorFen 40/100mg: study drug arm Atorvastatin 40mg and fenofibrate 100mg
- Atorvastatin 40mg: active control arm atorvastatin 40mg
- Fenofibrate 145mg: active control arm fenofibrate 145mg
Period: Overall Study
Arm/Group | LCP-AtorFen 40/100mg | Atorvastatin 40mg | Fenofibrate 145mg
Started | 73 | 74 | 73
Completed | 67 | 70 | 63
Not Completed | 6 | 4 | 10
Not completed — Protocol Violation | 6 | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCP-AtorFen 40/100mg | Atorvastatin 40mg | Fenofibrate 145mg | Total
Number analyzed (Participants) | 73 | 74 | 73 | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 73 | 74 | 73 | 220
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (10.74) | 56.3 (9.88) | 56.4 (10.58) | 55.9 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 39 | 33 | 105
  Male | 40 | 35 | 40 | 115
Region of Enrollment [Number; unit: participants]
  United States | 73 | 74 | 73 | 220

OUTCOME MEASURES:

1. Primary Outcome: Percent Changes From Baseline to End-of-treatment in Non-HDL Cholesterol, HDL Cholesterol, and Triglycerides by LCP-AtorFen Versus Atorvastatin Monotherapy
Description: Mean percent change from baseline to end-of-treatment (12 weeks) for non-HDL cholesterol and triglycerides and the mean percent change from baseline to end-of-treatment for HDL cholesterol for AtorFen 40/100mg fixed-dose combination tablet versus atorvastatin 40mg tablet.
Time Frame: baseline(randomization) to 12 weeks
Population: Modified intent-to-treat population consisted of all subjects randomized who had at least one dose of study drug and one post-baseline (randomization) assessment
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | LCP-AtorFen 40/100mg | Atorvastatin 40mg
Number analyzed (Participants) | 71 | 73
percent change from baseline
  non-HDL: number analyzed (Participants) | 67 | 70
  non-HDL | -44.8 (16.2) | -40.2 (17.3)
  triglycerides: number analyzed (Participants) | 67 | 70
  triglycerides | -49.1 (24.46) | -28.9 (32.25)
  HDL: number analyzed (Participants) | 67 | 70
  HDL | 19.7 (21.38) | 6.5 (18.77)

2. Secondary Outcome: Percent Changes From Baseline to End-of-treatment in Non-HDL, HDL and LDL Cholesterol by LCP-AtorFen Versus Fenofibrate Monotherapy
Description: Mean percent changes from baseline (Visit 3, Week 0) to end-of-treatment (Visit 6; Week 12) in non-HDL, HDL and LDL cholesterol by LCP-AtorFen versus fenofibrate monotherapy
Time Frame: baseline (week 0) to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | LCP-AtorFen 40/100mg | Fenofibrate 145mg
Number analyzed (Participants) | 71 | 73
percent change from baseline
  non-HDL: number analyzed (Participants) | 67 | 63
  non-HDL | -44.8 (16.2) | -16.1 (17.5)
  LDL: number analyzed (Participants) | 62 | 59
  LDL | -42.3 (20.01) | -13.9 (18.31)
  HDL: number analyzed (Participants) | 67 | 63
  HDL | 19.7 (21.38) | 18.2 (17.81)

ADVERSE EVENTS:
Description: For certain "Other (Not Including Serious) Adverse Events" some adverse events were monitored/assessed without regard to a specific adverse event term, and were therefore listed only by organ class.
Arm/Group | LCP-AtorFen 40/100mg | Atorvastatin 40mg | Fenofibrate 145mg
Serious Adverse Events (participants affected / at risk) | 1/73 | 0/74 | 2/73
Other Adverse Events (participants affected / at risk) | 43/73 | 49/74 | 48/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCP-AtorFen 40/100mg (N=73) | Atorvastatin 40mg (N=74) | Fenofibrate 145mg (N=73)
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCP-AtorFen 40/100mg (N=73) | Atorvastatin 40mg (N=74) | Fenofibrate 145mg (N=73)
Endocrine Disorders (any) (Endocrine disorders) | 0 | 2 | 0 — specific adverse event unknown
Gastrointestinal Disorders (any) (Gastrointestinal disorders) | 13 | 9 | 10
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 3 | 1 | 3
Gastro esophageal reflux diseases (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
General Disorders and Administration Site Conditions (General disorders) | 5 | 1 | 5
Fatigue (General disorders) | 2 | 0 | 3
Infections and Infestations (any) (Infections and infestations) | 10 | 18 | 13
Bacteriuria (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 4 | 8 | 2
Sinusitis (Infections and infestations) | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 2
Injury, Poisoning and Procedural Complications (any) (Injury, poisoning and procedural complications) | 3 | 2 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Investigations (any) (Investigations) | 13 | 11 | 13
Alanine aminotransferase increased (Investigations) | 3 | 5 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 4 | 2 | 2
Blood glucose increased (Investigations) | 2 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 2 | 0 | 5
Gamma- glutamyltransferase increased (Investigations) | 2 | 0 | 2
Liver function test abnormal (Investigations) | 2 | 0 | 1
Metabolism and Nutrition (any) (Metabolism and nutrition disorders) | 1 | 1 | 3
Musculoskeletal and Connective Tissue Disorders (any) (Musculoskeletal and connective tissue disorders) | 8 | 9 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neoplasms Benign, Malignant and Unspecified (any) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 — specific adverse event unknown
Nervous System Disorders (any) (Nervous system disorders) | 5 | 5 | 2
Headache (Nervous system disorders) | 1 | 2 | 0
Psychiatric Disorders (any) (Psychiatric disorders) | 0 | 1 | 2 — specific adverse event unknown
Renal and Urinary Disorders (any) (Renal and urinary disorders) | 0 | 2 | 3 — specific adverse event unknown
Reproductive System and Breast Disorders (any) (Reproductive system and breast disorders) | 1 | 1 | 2 — specific adverse event unknown
Respiratory, Thoracic and Mediastinal Disorders (any) (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Skin and Subcutaneous Tissue Disorders (any) (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Vascular Disorders (any) (Vascular disorders) | 3 | 2 | 2
Hypertension (Vascular disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual investigators may publish data arising from their own subjects. The Principal Investigator will provide the Sponsor with copies of written publications (including abstracts and posters) at least 60 days in advance of submission.